CLINICAL TRIAL: NCT04305197
Title: A Phase Ib/IIa Double-blind, Randomized, Placebo-controlled Study to Evaluate the Safety, Tolerance, Pharmacokinetics/ Pharmacodynamics(PK/PD) of ICP-022 in Patients With Mild and Moderate Systemic Lupus Erythematosus
Brief Title: A Study of ICP-022 in Patients With Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICP-CL-00109
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Mild to Moderate
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — orelabrutinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lower Dose (Experimental)
  Interventions: Drug: ICP-022
- Medium Dose (Experimental)
  Interventions: Drug: ICP-022
- Higher Dose (Experimental)
  Interventions: Drug: ICP-022
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: ICP-022 — Tablet, 50mg, once a day, oral, will be administered for 12 weeks in double-blind treatment period
  Other Names: Orelabrutinib
  Arms: Lower Dose
Drug: ICP-022 — Tablet, 80mg, once a day, oral, will be administered for 12 weeks in double-blind treatment period
  Other Names: Orelabrutinib
  Arms: Medium Dose
Drug: ICP-022 — Tablet, 100mg, once a day, oral, will be administered for 12 weeks in double-blind treatment period
  Other Names: Orelabrutinib
  Arms: Higher Dose
Drug: Placebos — Tablet, matched to ICP-022, once a day, oral, will be administered for 12 weeks in double-blind treatment period
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the Safety, Tolerability, PK/PD and preliminary Efficacy of ICP-022 in Subjects with Systemic Lupus Erythematosus (SLE)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 to 75
2. diagnosis of with SLE at least 6 months at screening visit
3. SLEDAE-2K≥5
4. Is receiving standard treatment for SLE and has been receiving treatment for at least 3 months.
5. At least one SLE activity manifestation (as assessed by SLEDAE-2K)

Exclusion Criteria:

1. Failure to comply with the requirements of the programme
2. A female or male partner who is pregnant or breastfeeding or who plans to become pregnant during the study period
3. Previously treated with a BTK inhibitor
4. Neuropsychiatric lupus (NPSLE)
5. Has other autoimmune diseases other than SLE

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Number of participants that experience Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 28 Days after the last dose of study drug
Number of Patients with Treatment-emergent Adverse Event(TEAEs) according to severity | Up to 28 Days after the last dose of study drug
Number of participants with clinically significant physical examination abnormalities | Up to 28 Days after the last dose of study drug
Number of participants with clinically significant vital signs abnormalities | Up to 28 Days after the last dose of study drug
Number of participants with clinically significant ECG abnormalities | Up to 28 Days after the last dose of study drug
Number of participants with clinically significant laboratory examination abnormalities | Up to 28 Days after the last dose of study drug

SECONDARY OUTCOMES:
Ratio of Patients With Response Based on Systemic Lupus Erythematosus Responder Index 4 (SRI-4) | 12 Weeks
Ratio of Patients With Response Based on Systemic Lupus Erythematosus Responder Index 6 (SRI-6) | 12 Weeks
Occupancy rate of Bruton Tyrosine Kinase(BTK) | 14 Days
Serum Immunoglobulin (Ig) level | 12 Weeks
Changes from Baseline in Ig levels | 12 Weeks
Changes from Baseline in C3 | 12 Weeks
Changes from Baseline in C4 | 12 Weeks
Changes from Baseline in serum dsDNA | 12 Weeks
Changes from Baseline in Anti-nuclear Antibodies | 12 Weeks
Changes from Baseline in Interferon-α(INF-α) level | 12 Weeks
  Changes from Baseline in cytokine levels
Changes from Baseline in Interleukin-6(IL-6) level | 12 Weeks
  Changes from Baseline in cytokine levels
Changes from Baseline in total B cell counts | 12 Weeks
Change from Baseline in Beffs count | 12 Weeks
Changes from baseline in Bregs count | 12 Weeks
Changes from Baseline in Bregs to Beffs ratio | 12 Weeks
Changes from Baseline in Erythrocyte Sedimentation Rate(ESR) | 12 Weeks
The plasma concentration-time curve | 14 Days

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, MD/PhD, Principal Investigator — Peking University People's Hospital
Locations (11):
- China (11):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University third hospital, Beijing, Beijing Municipality
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - University of Hong Kong Shenzhen Hospital, Shenzhen, Guangdong
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Gulou Hospital Affiliated to Medical College of Nanjing University, Nanjing, Jiangsu
  - Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No